CLINICAL TRIAL: NCT01108913
Title: Multi-center, Randomized, Double-blind, Placebo-controlled, Cross-over Phase II Study to Evaluate the Safety and Efficacy of Inhaled Bimosiamose for the Treatment of Patients With Moderate to Severe COPD
Brief Title: Study to Evaluate Safety and Efficacy of Inhaled Bimosiamose for the Treatment of Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revotar Biopharmaceuticals AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: R015
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — bimosiamose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bimosiamose (Active Comparator)
  Interventions: Drug: Bimosiamose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bimosiamose
  Arms: Bimosiamose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether inhalation of Bimosiamose is safe and effective in the treatment of patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal or sterile female patients with a history of moderate to severe COPD defined as Global Initiative for Chronic Obstructive Lung Disease (GOLD) II-III for at least 1 year
* At least 40 years of age
* Current smoker or ex-smoker with at least 10 pack-year smoking history (Ten pack-years is defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.)
* Postbronchodilator FEV1 between 30% and 80% predicted and FEV1/FVC ratio < 70%. Postbronchodilator refers to 30 min after inhalation of 400 µg Salbutamol. This criterion for FEV1 will have to be demonstrated after a washout period of at least 48 h during which no long acting anticholinergic medication (LAMA) or long acting β2-agonists (LABA) has been inhaled or a washout period of 6 h during which no short acting β2-agonists (SABA) or anticholinergic medication (SAMA) has been inhaled. For patients having been pretreated with an inhaled corticosteroid (ICS) and/or theophylline, this criterion needs to be demonstrated after a washout of at least 4 weeks.
* Able to produce sputum upon induction in a sufficient quality. This criterion will be checked by the responsible sputum lab prior to randomization of the patient.
* Time and ability to complete the study
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.

Exclusion Criteria:

* Patients with a history of chronic respiratory disorders other than COPD e.g. asthma, α1-Antitrypsin deficiency, mucoviscidosis, lung fibrosis
* Patients who experienced an exacerbation in the 4 weeks before the screening visit or between screening and randomization
* Patients who experienced an acute upper respiratory tract infection or broncho-pulmonary infection requiring antibiotic treatment during the 4 weeks before the screening visit or between screening and randomization
* Treatment with inhaled (ICS), topical or any systemic corticosteroids or theophylline within at least 4 weeks before the screening visit and throughout entire course of the study. Patients with ICS and/or theophylline treatment will undergo a washout of at least 4 weeks after signature of the informed consent and prior to the screening visit, where eligibility to enter the study will be assessed

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

PRIMARY OUTCOMES:
difference in absolute neutrophil cell counts and interleukin-8 in induced sputum between Bimosiamose and placebo treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Insaf - Respiratory Research Institute GmbH, Wiesbaden, Germany

REFERENCES:
- [Derived] Watz H, Bock D, Meyer M, Schierhorn K, Vollhardt K, Woischwill C, Pedersen F, Kirsten A, Beeh KM, Meyer-Sabellek W, Magnussen H, Beier J. Inhaled pan-selectin antagonist Bimosiamose attenuates airway inflammation in COPD. Pulm Pharmacol Ther. 2013 Apr;26(2):265-70. doi: 10.1016/j.pupt.2012.12.003. Epub 2012 Dec 17. PMID 23257347
- [Derived] Kirsten A, Watz H, Kretschmar G, Pedersen F, Bock D, Meyer-Sabellek W, Magnussen H. Efficacy of the pan-selectin antagonist Bimosiamose on ozone-induced airway inflammation in healthy subjects--a double blind, randomized, placebo-controlled, cross-over clinical trial. Pulm Pharmacol Ther. 2011 Oct;24(5):555-8. doi: 10.1016/j.pupt.2011.04.029. Epub 2011 Apr 14. PMID 21514398